CLINICAL TRIAL: NCT04227509
Title: A Randomized Phase II Study of CONsolidation PEmbrolizumab After Chemoradiotherapy in Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Consolidation Pembrolizumab After Chemoradiotherapy in Locally Advanced Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bhumsuk Keam, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CONPELAN
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients will be treated with pembrolizumab after concurrent chemoradiotherapy with cisplatin. Patients will be treated with up to 12 months (17 cycles) of pembrolizumab until disease progression or recurrence.
  Interventions: Drug: Pembrolizumab
- Placebo (Placebo Comparator): Patients will not be treated with pembrolizumab and will be treated with normal saline after concurrent chemoradiotherapy. Patients will be treated with up to 12 months (17 cycles) of pembrolizumab until disease progression or recurrence.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks.
  Arms: Experimental
Drug: Placebo — normal saline will be administered as a 30 minute IV infusion every 3 weeks.
  Arms: Placebo

SUMMARY:
Patients will be treated with pembrolizumab after concurrent chemoradiotherapy with cisplatin. Patients will be treated with up to 17 cycles (approximately 1 year) of pembrolizumab until disease progression or recurrence

DETAILED DESCRIPTION:
Phase II multi-center, randomized controlled trial of consolidation pembrolizumab after chemoradiotherapy in locally advanced nasopharyngeal carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically diagnosed nasopharyngeal carcinoma(NPC)

   1. WHO Type 2a, 2b nonkeratinizing, undifferentiated subtype
   2. Keratinizing subtype is excluded due to less associated with EBV infection
2. Stage II-IVB Locally advanced disease

   a. Stage II-IVB disease must confirmed by initial CT and/or MRI, PET CT at initial diagnosis according to the AJCC 8th edition
3. Prior Therapy

   1. Patients must have received curative radiotherapy (radiation dose ≥ 60Gy) and concurrent cisplatin (cumulative dose ≥ 200mg/m2)
   2. Induction chemotherapy followed by CCRT is permissible
   3. CCRT followed by adjuvant FP is permissible
   4. Patients must have recovered Gr2 or less than Gr2 from all acute, reversible toxic effects from chemotherapy and radiotherapy (excluding alopecia)
4. Age 19 or more than 19 years old
5. The patient must have an ECOG performance status of 0, 1
6. Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
7. patient with the willingness to comply with the study protocol during the study period and capable of complying with it
8. A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages. Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrolment in the trial to document their willingness to participate.
9. Have adequate organ function as defined in the following . Specimens must be collected within 10 days prior to the start of study treatment.

Hematological Absolute neutrophil count (ANC) ≥1500/µL Platelets ≥100 000/µL Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La Renal Creatinine ≤1.5 × ULN OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN Hepatic Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)

Exclusion Criteria:

1. Participants are excluded for patients with a history of other malignancies

   a. except: adequately treated non-melanoma skin cancer, early gastric cancer, curatively treated in-situ cancer, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years following the end of treatment and, which, in the opinion of the treating physician, do not have a substantial risk of recurrence of the prior malignancy.
2. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

   a. Patients with Grave's disease and/or psoriasis not requiring systemic therapy within the last two years from randomization are not excluded.
3. History of primary immunodeficiency, history of organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of randomization or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy.

   1. Intranasal/inhaled corticosteroids or systemic steroids that do not to exceed 10 mg/day of prednisone or equivalent dose of an alternative corticosteroid are permissible.
   2. pneumonitis that has required a course of oral steroids to assist with recovery, or a history of interstitial lung disease
4. History of diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal carcinomatosis which are known risks factors for bowel perforation
5. Live attenuated vaccination administered within 30 days prior to randomization.
6. History of severe hypersensitivity (≥Grade 3) to pembrolizumab
7. Mean QTc correction > 470msec in screening ECG measured using standard institutional method or history of familial long QT syndrome.
8. Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects). Patients with a significant cardiac history, even if controlled, should have a LVEF > 50% within 12 weeks prior to randomization.
9. Concurrent treatment with other investigational drugs or anti-cancer therapy.
10. Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol. This includes but is not limited to:

    1. known active tuberculosis (inactive tuberculosis or tuberculosis scar are allowed)
    2. known acute hepatitis B or C by serological evaluation (inactive healthy HBsAg carriers treated with pre-emptive anti-viral agents were allowed)
    3. known human immunodeficiency virus infection.
11. Active symptomatic central nervous system (CNS) metastases that the disease also has to have demonstrable stability with no evidence of growth and has not required recent steroid use and/or carcinomatous meningitis
12. Active infection requiring therapy
13. Symptomatic ascites or pleural effusion
14. Pregnant or lactating women. Women of childbearing potential must have a urine pregnancy test proven negative within 14 days prior to randomization. Men and women of child-bearing potential must agree to use adequate contraception as described in protocol
15. Prior organ transplant or allogeniec bone marrow transplant regardless of whether immunosuppressive therapy has been used in the past

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
3-year progression-free survival (PFS) rate | 3 years after the first date of treatment
  The percentage of patients who have not experienced disease progression or death from any cause within 3 years from the start of treatment.

SECONDARY OUTCOMES:
Objective Response rate (RR) | 1 year after the first date of treatment
  The percentage of patients who are either CR or PR within 3 years from the start of treatment.
Overall survival (OS) | 3 years after the first date of treatment
  The duration from the first date of treatment to the date of death from any cause or follow-up
median Progression-free survival (PFS) | 3 years after the first date of treatment
  The time at which half of the patients in a study have experienced disease progression or death, and half have not.

CONTACTS AND LOCATIONS:
Overall Officials: Bhumsuk Keam, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Department of Internal Medicine, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No